CLINICAL TRIAL: NCT00672269
Title: A Pilot Study to Investigate Germ-Line MEN1 and SDHD Gene Mutation in Familial Cases of Carcinoid Cancer
Brief Title: Study Investigating MEN1 and SDHD in Familial Carcinoid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rutgers University (Other)
Responsible Party: Nancy Gardner PhD Principal Investigator, Rutgers University
Other Study IDs: 08-451
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoid Neuroendocrine Cancer
Keywords: carcinoid; family members; familial; tumors; cancer
MeSH Terms: conditions — Carcinoid Tumor; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: a small sample of 2 tubes (2 - 4 teaspoons, or 20 ml). One tube will be used to prepare the DNA (your genetic material) for the test. The other would be used for further gene evaluation. The DNA will be stored with Rutgers University Cell and DNA Repository (RUCDR).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Families with carcinoid in multiple family members

SUMMARY:
There is a high incidence among the first degree relatives of the carcinoid patients, indicating the involvement of genetic components in its initiation and pathogenesis.

DETAILED DESCRIPTION:
This proposed pilot study will conduct detailed interviews into the medical, environmental, and family histories and to collect blood specimen to obtain DNA. The Blood specimen and DNA will be processed by the Rutgers University Cell and DNA Repository (RUCDR) to rule out Familial Multiple Endocrine Neoplasia (MEN 1), and succinate dehydrogenase complex, subunit D (SDHD), gene inactivation thought to be associated with different types of carcinoid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years
2. More than one ,member of a family with a history of biopsy confirmed carcinoid tumor
3. English speaking
4. Mentally and emotionally capable of answering questions
5. Willing and available for study participation
6. At least one other family member with carcinoid tumor

Exclusion Criteria:

1. If you are under the age of 18 years,
2. If you are unable to understand or unable to provide informed consent,
3. If you have a psychological condition (i.e. depression, anxiety disorder, substance abuse, etc.) which might cause you significant problems in dealing with test results.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with carcinoid cancer that report to have a first-degree family member also with carcinoid tumor
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Mutations in MEN1 and SDHD genes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Gardner, PhD, Principal Investigator — Rutgers University; Changshun Shao, PhD, Principal Investigator — Rutgers University
Locations (1):
- Busch Campus of Rutgers University, Human Genetics Institute, Piscataway, New Jersey, United States